CLINICAL TRIAL: NCT00931086
Title: An Expanded Access Trial of Belimumab Antibody (Monoclonal Anti-BLyS Antibody) in Patients With Rheumatoid Arthritis (RA) Who Were Previously Treated Under HGS Protocol LBRA99
Brief Title: Expanded Access Trial of Belimumab Antibody in RA Patients Who Were Previously Treated Under HGS Protocol LBRA99
Acronym: LBRA99
Status: No longer available | Type: Expanded Access
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Other Study IDs: HGS1006-C1089
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — belimumab

INTERVENTIONS:
Drug: belimumab — IV 10mg/kg q28days
  Other Names: BENLYSTA™ (belimumab); LymphoStat-B™

SUMMARY:
An expanded access trial of belimumab for named patients who participated in LBRA99.

DETAILED DESCRIPTION:
An expanded access trial of belimumab for named patients with Rheumatoid Arthritis (RA) who have experienced continued benefit under HGS Protocol LBRA99.

ELIGIBILITY:
Inclusion Criteria:

1. Have in the clinical judgment of the investigator, experienced significant clinical benefit while on belimumab treatment in the HGS Protocol LBRA99.
2. Over the course of the study and for 60 days after the last dose of study agent, any woman with an intact uterus who is not post-menopausal must agree to practice a medically accepted method of contraception.
3. Over the course of the study and for 60 days after the last dose of study agent, all men must agree to practice a medically accepted method of contraception.
4. Have the ability to understand the requirements of this study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the required study visits.

Exclusion Criteria:

1. Had not been previously treated with belimumab in LBRA99 or were discontinued from treatment prior to HGS' decision to terminate LBRA99.
2. Had clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to RA (ie, cardiovascular, pulmonary, anemia, gastrointestinal, hepatic, renal, neurological, cancer or infectious diseases) that could, in the opinion of the principal investigator, put the patient at undue risk.
3. Are a pregnant female or nursing mother.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Rheumatology Associates of Central Florida, Orlando, Florida, United States